CLINICAL TRIAL: NCT06388902
Title: A Phase I Clinical Study of the Safety, Tolerability and Efficacy of BR115 for Injection in Patients With Advanced Solid Malignancies
Brief Title: A Phase I Study of BR115 for Injection Alone in Subjects With Advanced Solid Malignancies
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to drug stability and global interests, it is currently in a suspended state.
Sponsor: BioRay Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR115-101
Record Dates: First submitted 2024-01-31; First posted 2024-04-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Malignancies
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BR115 (Experimental)
  Interventions: Drug: BR115 for injection

INTERVENTIONS:
Drug: BR115 for injection — BR115 for injection will be administered by subcutaneous injection, two doses at the first week of treatment, followed by once per week until intolerable toxicity, disease progression, pregnancy, withdrawal of informed consent, death, study discontinuation or withdrawal from the study. The dose of each administration will be calculated based on the weight measured prior to such administration. The dosing regimen (dosing frequency and interval) for subsequent study may be adjusted based on prior data.

SUMMARY:
This is a Phase I, multicenter, open-label, single-arm and first-in-human clinical study of BR115 for injection. The study objectives are to evaluate the safety, tolerability, pharmacokinetic profile, anti-tumor activity and immunogenicity of BR115 for injection in patients with advanced solid malignancies.

Patients will receive two doses at the first week of treatment, followed by once per week until intolerable toxicity, disease progression, pregnancy, withdrawal of informed consent, death, study discontinuation, or withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

* (1) Subjects who voluntarily sign the informed consent form, understand the nature, objectives, and procedure of the study and are able to complete the study according to the protocol; (2) ≥18 years of age (based on the date of signing the informed consent form); (3) In Phase Ia: patients must have advanced solid tumors confirmed by histopathology and/or cytology, the expression of HER2 was confirmed by the laboratory（IHC3+、or IHC2+ and FISH+、or IHC2+ and ISH-、or IHC1+）who have failed to respond to standard-of-care (disease progression after treatment) or who could not tolerate standard-of-care, or who could not obtain effective standard-of-care or for whom there was no effective standard-of-care available; (Note: the patient population and inclusion criteria in phase Ib will be determined according to the data of phase Ia); (4) According to RECIST v1.1 (Response Evaluation Criteria in Solid Tumors), there is at least 1 measurable lesion; (5) Eastern Cooperative Oncology Group (ECOG) Status 0 to 1; (6) Adequate organ and bone marrow function (no treatment with cells, growth factors, or transfusions within 14 days prior to the first administration), as defined below:

  1. Hematology: absolute neutrophil count (ANC) ≥ 1.0 × 109/L, platelet count (PLT) ≥ 100 × 109/L, hemoglobin (HGB) ≥ 80 g/L，the lymphocyte count is normal ≥ 0.8 × 109/L;
  2. Liver function: serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN) (except for subjects with Gilbert syndrome, TBIL ≤ 2 × ULN in patients with liver cancer or liver metastases), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (in patients with liver cancer or liver metastases, ALT or AST ≤ 5 × ULN);
  3. Renal function: creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance (CrCL) (based on Cockcroft-Gault equation) ≥ 60 mL/min;
  4. Lung function：Vital capacity and forced expiratory volume in the first second (FEV1) were > 65% of the normal predicted value, and diffusion capacity was > 55% of the normal predicted value； (7) Expected survival ≥ 12 weeks; (8) Female subjects with fertility potential must test negative for serum human chorionic gonadotropin (HCG) before they are enrolled in the study. Female subjects with fertility potential or male subjects who have a female partner must agree to maintain no pregnancy plan and take effective contraceptive measures such as condoms from the signing of ICF to 6 months after the last dose of study drug; females are considered fertile from menarche to menopause (at least 12 months without menstruation) unless they are permanently infertile (through hysterectomy, bilateral salpingectomy, or bilateral oophorectomy).

Exclusion Criteria:

* (1) Subjects who have previous hypersensitivity to BR115 or known hypersensitivity to any component or excipient of the study drug; (2) Subjects who have any active infections, including bacterial, viral, fungal, mycobacterial, parasitic, or other infections (excluding onychomycosis) , were present at the time of first administration; (3) Subjects who have previous or current presence of two or more primary tumors (excluding cured cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma of the skin, and other tumors that have been stable for more than 5 years after treatment); (4) Subjects who have symptoms of active central nervous system metastases； (5) Subjects with serious cardiovascular and cerebrovascular diseases and lung diseases, including but not limited to:

  1. Stroke, intracranial hemorrhage, unstable angina pectoris, congestive heart failure (NYHA class III-IV), myocardial infarction, severe arrhythmias (such as sustained ventricular tachycardia and ventricular fibrillation), congenital long QT syndrome, torsade de pointes, and symptomatic pulmonary embolism within 6 months before enrollment;
  2. Uncontrolled hypertension (at least 2 consecutive measurements of systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg);
  3. Echocardiogram (ECHO) or multigated acquisition scan (MUGA) shows left ventricular ejection fraction (LVEF) < 50%;
  4. During the screening period, the mean corrected (by Fridercia's formula) QT interval on three consecutive electrocardiograms is prolonged (> 450 ms in males and > 470 ms in females);
  5. Subjects who have interstitial lung diseases, severe impaired lung function, severe pulmonary fibrosis, radiation pneumonitis, and other lung diseases assessed by the investigator as clinically significant; (6) (6) Gastrointestinal disorders considered clinically significant by the investigators (e.g. , including liver disease, bleeding, inflammation, obstruction, intestinal obstruction, grade 1 diarrhea, jaundice, intestinal paralysis, malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, or partial intestinal obstruction); (7) Subjects who have undergone major surgery within 4 weeks prior to the first dose of study drug or are expected to be performed during the study; (8) Subjects who have a history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; (9) Subjects who have used strong inhibitors or substrates of CYP3A4 and/or Pgp within 4 weeks before the first dosing or within 5 half-lives of the used drug (whichever is shorter), or who have received anti-tumor therapy or participated in other clinical studies and used other study drugs, including chemotherapy, targeted therapy, immunotherapy, biotherapy (tumor vaccines, cytokines, or growth factors for cancer control), etc.; or who have received prepared slices of Chinese crude drugs or Chinese patent medicines as anti-tumor treatment within 1 week before the first dose of study drug; (10) Systemic immunosuppressants/agonists (drugs with longer half-lives) , such as PD1, CTLA4,41BB, were used within 4 half-lives before the first administration; (11) Subjects who have received radiation therapy, including abdominal palliative stereotactic radiotherapy, within 4 weeks prior to the first dose of study drug (non-abdominal palliative stereotactic radiotherapy within 2 weeks prior to the first dose); (12) Toxicity of previous antineoplastic therapy does not resolve to grade ≤ 1 as defined by NCI-CTCAE v5.0 (except for asymptomatic abnormal laboratory findings considered by the investigator, such as elevated ALP, hyperuricemia, elevated blood glucose, etc.; except for toxicity with no safety risk determined by the investigator , such as alopecia, pigmentation, etc.); (13) Subjects who have been vaccinated with a live vaccine within 4 weeks before the first dose, or who intend to be vaccinated with a live vaccine during the study; (14) Subjects who have received more than 1 week of treatment with systemic corticosteroids (methylprednisolone > 10 mg/day or an equivalent dose of other similar drug) within 2 weeks prior to the first dose of study drug; (15) Subjects who have used immunosuppressants within 2 weeks prior to the first dose or once had active autoimmune diseases or had a prior history of autoimmune diseases; (16) Subjects who test positive for Hepatitis B surface antigen (HBsAg) with HBV DNA beyond the normal range; or subjects who test positive for hepatitis B core antibody with HBV DNA beyond the upper limit of normal, but do not agree to regular DNA testing during treatment and follow-up, or do not agree to receive antiviral therapy; subjects who test positive for hepatitis C virus (HCV) antibody and HCV RNA; subjects who are seropositive for human immunodeficiency virus (HIV); subjects who have syphilis and need to receive systemic treatment; (17) Subjects who are pregnant or breastfeeding; (18) Subjects who are not eligible for enrollment by the investigator's assessment.;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent Adverse Events Following Treatment With BR115 | From date of randomization until the date of first documented progression or date of death from any cause or date of documented unacceptable toxicity , assessed up to 24 months
  Adverse events (AEs) will be assigned severity grades based on Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. A treatment-emergent adverse event (TEAE) is defined as an AE that occurred, having been absent before the first dose of study drug.

SECONDARY OUTCOMES:
Objective Response Rate | From date of randomization until the date of first documented progression or date of death from any cause or date of documented unacceptable toxicity , assessed up to 24 months
  Defined as participants (who will achieve CR and PR) will be assessed by the investigator based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR is defined as a disappearance of all target lesions and PR is defined as at least a 30% decrease in the sum of diameters of target lesions.
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause or date of documented unacceptable toxicity , assessed up to 24 months
  TProgression-free survival (PFS) by independent central review is defined as the time from the date of enrollment to the earlier of the dates of the first objective documentation of disease progression (as per RECIST v1.1) or death due to any cause
Overall survival (OS) | Baseline up to 2 years.
  Overall survival (OS) by independent central review is defined as the time interval from the date of enrollment to the date of death from any cause.
Disease control rate (DCR) | From date of randomization until the date of first documented progression or date of death from any cause or date of documented unacceptable toxicity , assessed up to 24 months
  Disease control rate (DCR; defined as participants who will achieve CR, PR, and SD) will be assessed by the investigator based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR is defined as a disappearance of all target lesions, PR is defined as at least a 30% decrease in the sum of diameters of target lesions, and SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD defined as at least a 20% increase in the sum of diameters of target lesions.
Duration of response (DOR). | From date of randomization until the date of first documented progression or date of death from any cause or date of documented unacceptable toxicity , assessed up to 24 months
  Duration of response (DoR) by independent central review is defined as the time between the date of the first complete response (CR) or partial response (PR) until the date of the first documentation of progressive disease (PD) or death due to any cause. CR is defined as a disappearance of all target lesions, PR as at least a 30% decrease in the sum of diameters of target lesions, and PD as at least a 20% increase in the sum of diameters of target lesions.
Pharmacokinetic Parameter Maximum Serum Concentration (Cmax) | Cycle 1, Day1，Days 4 and Days 8: 0 hours, 4 hours, 8 hours; 24 hours; Days 8:72 hours; Days 15: 0 hours; cycle2: Days 1,Days 8,Days 15; cycle3：Days1: 0 hours,4 hours,8 hours ,24 hours,72 hours ,Days 8;Cycle 4-n: Day 1: 0hours (each cycle is 21 days)
  Cmax of BR115 will be assessed.
Pharmacokinetic Parameter Area Under the Concentration-time Curve (AUC) | Cycle 1, Day1，Days 4 and Days 8: 0 hours, 4 hours, 8 hours; 24 hours; Days 8:72 hours; Days 15: 0 hours; cycle2: Days 1,Days 8,Days 15; cycle3：Days1: 0 hours,4 hours,8 hours ,24 hours,72 hours ,Days 8;Cycle 4-n: Day 1: 0hours (each cycle is 21 days)
  Area under the concentration-time curve of BR115 will be assessed
The anti-drug antibody (ADA) | Cycle 1, Day1: before first infusion; Days 8: before third infusion; Days 15: before fourth infusion; Cycle 2~n, Day 1: before first infusion ; (each cycle is 21 days)
  The anti-drug antibody (ADA) of BR115 will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No